CLINICAL TRIAL: NCT01041924
Title: Dynamic Carbon Dioxide Administration for Central Sleep Apnoea in Heart Failure
Brief Title: Dynamic Carbon Dioxide (CO2) Administration for Sleep Apnoea
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Dr Darrel P Francis, Imperial College
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: FS/04/079
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Last update posted 2010-01-05 (Estimated); Status verified 2010-01

CONDITIONS: Sleep Apnea, Central
Keywords: Sleep apnea; Periodic breathing; Heart Failure
MeSH Terms: conditions — Sleep Apnea, Central; Sleep Apnea Syndromes; Heart Failure | interventions — Carbon Dioxide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Carbon dioxide — 2% inhaled CO2 for up to 8 hours.
Other: Carbon dioxide — Up to a maximum of 2% CO2, only delivered for a maximum of up to 20 seconds per 60 seconds for 8 hours

SUMMARY:
Normally breathing is controlled by a reflex that responds to the levels of carbon dioxide (CO2) in the blood. In heart failure, where the heart muscle is damaged and therefore does not pump as well, this reflex is exaggerated. The result is a vicious circle: blood CO2 levels fluctuate wildly and as a result breathing also fluctuates with patients hyperventilating at times and briefly stopping breathing at others. During sleep this is called central sleep apnoea (CSA).

Patients with CSA wake up throughout the night and whilst some patients are oblivious to this, others are consciously breathless and many patients are tired during the day and feel unable to perform their daily activities.

As part of the body's stress response to the erratic pattern of breathing, both blood pressure and heart rate may rise to a level that is harmful in a failing heart, exacerbating the underlying heart failure. Indeed patients who demonstrate this CSA die sooner than those who have heart failure and stable breathing.

There are no proven specific therapies for CSA that stabilise breathing, improve sleep quality, and prolong life. We have designed a system which delivers very small doses of CO2, when the blood level of CO2 is predicted to be low. During short daytime recordings, using this system, we have demonstrated that it is possible to stabilise the body's CO2 levels.

We aim to test what happens when CO2 is given overnight whilst the patient is sleeping to see whether we can stabilise their breathing over longer durations and whether sleep quality could be improved so that patients are less tired during the day. In addition, we would like to measure whether the stress response is lessened if the breathing is successfully stabilised.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 to 79 years of age who have New York Heart Association (NYHA) functional class I through IV heart failure due to ischemic, hypertensive, or idiopathic dilated cardiomyopathy and whose condition had been stabilized by means of optimal medical therapy for at least one month;
* An LVEF of less than 40% and central sleep apnea, defined as 15 or more episodes of apnea and hypopnea per hour of sleep, more than 50 percent of which are determined to be central rather than obstructive.

Exclusion Criteria:

* Pregnancy,
* Myocardial infarction,
* Unstable angina or cardiac surgery within the previous three months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-10 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Extent of respiratory instability | over 8 hours
Arousals | over 8 hours

SECONDARY OUTCOMES:
End-tidal CO2 | per breath
24 hour urinary catecholamines | per 24 hours
Mean heart rate | per 1 s
Number of ectopic heart beats | per 8 hours
Mean blood pressure | every 9 hours
Mean Ventilation | every 1 second

CONTACTS AND LOCATIONS:
Overall Officials: Darrel P Francis, MD, Principal Investigator — Imperial College London
Locations (2):
- Foundation G. Monasterio, Pisa, Pisa, Italy
- Imperial NHS Trust, London, London, United Kingdom

REFERENCES:
- See also: mathematical modelling work — http://www.ncbi.nlm.nih.gov/pubmed/19628721?itool=EntrezSystem2.PEntrez.Pubmed.Pubmed_ResultsPanel.Pubmed_RVDocSum&ordinalpos=2